CLINICAL TRIAL: NCT02031861
Title: Random, Open Label, Active Comparator-controlled Parallel Study to Evaluate the Efficacy of Nifedipine Controlled-released Tablets (Xin Ran) in Patients With Mild to Moderate Essential Hypertension
Brief Title: Efficacy Study of Nifedipine Controlled-Release Tablets (Xin Ran) to Treat Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Shyndec Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-004PIV
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2014-04

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nifedipine CR tablets (Xin Ran) (Experimental): Subjects will take a nifedipine controlled-release tablet (30 mg, Xin Ran) orally in every morning for a 12-week treatment period.
  Interventions: Drug: nifedipine CR tablets (Xin Ran)
- nifedipine CR tablets (Adalat) (Active Comparator): Subjects will take a nifedipine controlled-release tablet (30 mg, Adalat) orally in every morning for a 12-week treatment period.
  Interventions: Drug: nifedipine CR tablets (Adalat)

INTERVENTIONS:
Drug: nifedipine CR tablets (Xin Ran)
  Arms: nifedipine CR tablets (Xin Ran)
Drug: nifedipine CR tablets (Adalat)
  Arms: nifedipine CR tablets (Adalat)

SUMMARY:
The purpose of this study is to compare nifedipine controlled-release (CR) tablets (Xin Ran) with nifedipine controlled-release tablets (Adalat）in the treatment of mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and must sign informed consent form
* Mild to moderate essential hypertension (SBP 140-179 mmHg and/or DBP 90-109 mmHg)
* Average DBP measured by 24-hour ambulatory blood pressure monitoring (ABPM) ≥80 mmHg

Exclusion Criteria:

* Secondary hypertension and malignant hypertension
* Pregnant or nursing women, or patients that cannot guarantee to take effective contraception measures
* Baseline SBP≥180 mmHg or DBP≥110 mmHg, or patients with cerebral, cardiac or renal complications
* Have following complications: cerebrovascular accident within 6 months, myocardial infarction or cardiac failure, macroaneurysm or dissecting aneurysm, definite angina, A-V block of grade 2 or higher, sick sinus syndrome, atrial fibrillation or other malignant arrhythmia
* Clinical significant diseases of heart, lung, liver, kidney and hematologic system or malignant tumors, HIV infection, uncontrolled diabetes (fasting blood glucose ≥7.0 mmol/L, 2-hour postprandial blood glucose ≥7.8 mmol/L)
* Kock pouch
* Sever gastrointestinal stenosis
* Abnormal laboratory values with clinical significance, including serum potassium <3.5 or >5.5 mmol/L, glutamic-pyruvic transaminase (ALT) or glutamic oxalacetic transaminase (AST) >2-fold upper limit of normal (ULN), Cr >ULN
* Uric acid >ULN with the diagnosis of gout
* Gastrointestinal abnormalities or surgery that may interfere with drug absorption
* Hyperthyroidism or hypothyroidism
* Allergic to any ingredient or metabolite of investigational drug or drugs of similar structure
* Heavy smokers (>25 cigarettes every day), alcoholics (>250 ml liquor every day), drug addicts
* Psychological diseases, acrasia, cannot express explicitly
* Patients whose mood may be affected by variations in blood pressure, which in turn increases blood pressure
* Anxiety disorders, depression or cannot follow study protocol
* BMI >30
* Night shift, irregular sleep patterns or insomnia
* participate in other clinical trials within 3 months
* other conditions that investigators consider unsuitable for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change in morning blood pressure surge from baseline | 12 weeks
change in central systolic blood pressure, central diastolic blood pressure, central pulse pressure and augmentation index from baseline | 12 weeks

SECONDARY OUTCOMES:
change in morning blood pressure from baseline | 12 weeks
T/P ratio | 12 weeks
average reduction in systolic blood pressure from 18 to 24 hours after administration | 12 weeks
average reduction in diastolic blood pressure from 18 to 24 hours after administration | 12 weeks
smoothness index | 12 weeks
change in morning blood pressure surge from baseline | 8 weeks
change in central systolic blood pressure, central diastolic blood pressure, central pulse pressure and augmentation index from baseline | 8 weeks
change in morning blood pressure from baseline | 8 weeks
T/P ratio | 8 weeks
average reduction in systolic blood pressure from 18 to 24 hours after administration | 8 weeks
average reduction in diastolic blood pressure from 18 to 24 hours after administration | 8 weeks
smoothness index | 8 weeks
change in systolic blood pressure (SBP) from baseline | 12 weeks
change in diastolic blood pressure (DBP) from baseline | 12 weeks

OTHER OUTCOMES:
clinical laboratory test and adverse event | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pingjin Gao, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University Medical School
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University Medical School, Shanghai, Shanghai Municipality, China